CLINICAL TRIAL: NCT06039761
Title: Randomized Study Comparing the Combination Intraperitoneal Local Anesthetics, Maneuvers Alveolar Recruitment and Abdominal Compression Compared to Passive Exsufflation of the Pneumoperitoneum in the Prevention of Pain Shoulders After Laparoscopic Surgery
Brief Title: Randomized Study in the Prevention of Pain Shoulders After Laparoscopic Surgery
Acronym: POPPLaS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GCS Ramsay Santé pour l'Enseignement et la Recherche (Other)
Collaborators: Euraxi Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-A01281-44
Record Dates: First submitted 2023-09-08; First posted 2023-09-15 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Digestion

STUDY DESIGN:
Intervention Model Description: Study patients will be divided into 2 arms (1:1) and will benefit from one of the following procedures:
  * Arm A (experimental): Overall procedure = standard procedure + local intraperitoneal anesthetics + alveolar recruitment maneuver + abdominal compression maneuver.
  * Arm B (control): Standard procedure.
Who Masked: Participant
Masking Description: The patient will be blinded to the result of the randomization, unlike the investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- local intraperitoneal anesthetics + alveolar recruitment maneuver + abdominal compression maneuver (Experimental): Overall Procedure : The specific interventions are carried out at the end of the surgical intervention and include the use of intraperitoneal local anesthetics insufflated by the surgeon, the alveolar recruitment maneuver carried out by the anesthetist and that of abdominal compression carried out by the surgeon.
  Interventions: Procedure: Digestive or gynecological surgery by laparoscopy
- Standard Procedure (Active Comparator): Standard Procedure : Digestive or gynecological surgery by laparoscopy with a Transversus abdominis plane block before the incision and systematic standardized multimodal analgesia.
  Interventions: Procedure: Digestive or gynecological surgery by laparoscopy

INTERVENTIONS:
Procedure: Digestive or gynecological surgery by laparoscopy — Digestive or gynecological surgery by laparoscopy with a Transversus abdominis plane block before the incision and systematic standardized multimodal analgesia

SUMMARY:
The purpose of this study is to assess shoulder pain at rest (average over the last 24 hours) assessed by visual analogue scale from 0 to 100mm on Day 1.

DETAILED DESCRIPTION:
This is an interventional, comparative, controlled, randomized, single-blind study (the patient will be blinded to the result of the randomization, unlike the investigator) and single-center.

Comparative prospective cohort study of laparoscopic surgery with the addition of specific non-surgical interventions aimed at preventing postoperative shoulder pain (use of local intraperitoneal anesthetics, alveolar recruitment maneuver and compression maneuver abdominal) versus without specific interventions aimed at preventing post-operative shoulder pain.

All patients will benefit from Transversus Abdominis Plane block with multimodal analgesia provided in the usual setting of laparoscopic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Celiosurgery including a Transversus Abdominis Plane block with multimodal analgesia;
* Planned laparoscopic surgery for gallbladder, inguinal hernia, umbilical hernia, incisional hernia repair, adnexectomy, oophorectomy, endometriosis, tube ligation;
* Affiliation to the social security scheme;
* Signed informed consent

Exclusion Criteria:

* Celiosurgery such as colectomy, bariatric surgery, hysterectomy, prostatectomy, nephrectomy;
* Surgical emergency;
* History of chronic obstructive pulmonary disease;
* Weight less than 50 kg;
* Consumption of preoperative opioids;
* Antidepressant treatment and/or anxiolytic treatment;
* Conversion by laparotomy;
* Intraperitoneal sepsis;
* Major intraoperative complication (hemorrhage, anaphylaxis, etc.);
* Other surgical or medical interventions planned during the study;
* Patient participating in another clinical trial, or during a period of exclusion from another clinical trial;
* Inability to understand information related to the study;
* Woman who is pregnant or likely to be pregnant (of childbearing age, without effective contraception) or currently breastfeeding;
* Patient deprived of liberty or under guardianship or curatorship or unable to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2023-12-13 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Shoulder pain at rest assessed by visual analog scale | 1 day
  Shoulder pain at rest (average over the last 24 hours) assessed by visual analog scale from 0 to 100mm.
  ANCOVA (Analysis of Covariance) analysis will be applied to compare the mean shoulder pain visual analog scal (0 to 100 mm) between the groups, adjusted to the baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Privé Dijon Bourgogne, Dijon, France